CLINICAL TRIAL: NCT03016442
Title: Dinoprostone Vaginal Insert Versus Double Balloon Catheter for Preinduction Cervical Ripening
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Gonca Yetkin Yildirim, MD, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KanuniSSTRH -3
Record Dates: First submitted 2017-01-08; First posted 2017-01-10 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2016-11

CONDITIONS: Labor Induction
Keywords: Double balloon catheter; Dinoprostone; Labor induction
MeSH Terms: interventions — Dinoprostone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cook double balloon catheter (Experimental): A double- balloon catheter (Cook Cervical Ripener Balloon,Cook OB/GYN,Spencer IN) is inserted into cervical canal under direct visualisation during a sterile speculum examination İt is placed for 12 hours
  Interventions: Device: Cook Double Balloon Catheter
- Dinoprostone (Active Comparator): 10 mg of dinoprostone in a hydrogel insert is placed high in the vaginal fornix. İt is placed for 12 hours.It is a controlled release formulation which has been found to release dinoprostone in vivo at a rate of approximately 0.3 mg/hr.
  Interventions: Drug: Dinoprostone

INTERVENTIONS:
Device: Cook Double Balloon Catheter — A double- balloon catheter (Cook Cervical Ripener Balloon,Cook OB/GYN,Spencer IN) is inserted into cervical canal under direct visualisation during a sterile speculum examination.İt is placed for 12 hours
  Other Names: The Obstetric Cook Double Balloon Catheter
  Arms: Cook double balloon catheter
Drug: Dinoprostone — 10 mg of dinoprostone in a hydrogel insert is placed high in the vaginal fornix. İt is placed for 12 hours.It is a controlled release formulation which has been found to release dinoprostone in vivo at a rate of approximately 0.3 mg/hr.
  Other Names: Dinoprostone vaginal insert
  Arms: Dinoprostone

SUMMARY:
Effıcacy of dinoprostone vaginal insert versus double- balloon catheter among women in the induction of labor

DETAILED DESCRIPTION:
The study will be conducted in the Department of Obstetrics and Gynecology at Kanuni Sultan Süleyman Education and Research Hospital ,İstanbul, Turkey, with approval of the local institutional review board. All the participants will give informed consent before beginning of the study. Women who agree to participate will be first stratified into nulliparous and multiparous groups. Randomisation will be carried out by using sealed opaque envelopes with a piece of paper inside marked 'PGE2 vaginal insert' or 'Double-balloon catheter'. Envelopes will be prepared in blocks of 20 (10 PGE2 vaginal insert and 10 double-balloon catheters) for each stratified group. Envelopes will be then shuffled and placed in boxes marked 'nulliparous' and 'multiparous'. The investigator is not blinded to the allocation procedure. The allocated envelope will be opened by the clinician performing the initial vaginal examination just prior to that examination.

In the group assigned to mechanical ripening , a double- balloon catheter (Cook Cervical Ripener Balloon,Cook OB/GYN,Spencer IN) is inserted into cervical canal under direct visualisation during a sterile speculum examination. Once both balloon enter the cervical canal, the first balloon is filled with 40 ml saline above the level of the internal os. The second (vaginal) balloon is the inflated with 20 ml of saline.Then both of them are filled with 60 ml of saline. The external end of the device is taped without traction to the medial aspect of the woman's thigh. After completion of the device placement, patients undergo continous fetal heart rate monitoring for 30 min then are allowed to ambulate.The double ballon is placed for 12 hours .

In the group randomly assigned to vaginal insert is placed high in the vaginal fornix, the patients are monitored at least 1 hour for fetal heart rate and uterine activity and they are allowed to ambulate.

After 12 hours oxytocin isadministered using a standard dose regimen to all patients.

Primary and secondary outcomes are measured.

ELIGIBILITY:
Inclusion Criteria:

* Eligible women have obstetric or medical indications for labor induction with intact membranes
* singleton pregnancies,
* vertex presentations
* low Bishop scores ≤6
* gestational age ≥34 w
* reassuring fetal heart tracing on admission.

Exclusion Criteria:

* Exclusion criteria are placenta previa
* unexplained vaginal bleeding
* nonvertex presentation
* intrauterine fetal death
* prior cesarean delivery
* any scarred uterus
* any other contraindications for vaginal delivery.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Vaginal delivery after initiation of ripening within 24 hours | 24 hours

SECONDARY OUTCOMES:
Occurence of cesarean section | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Süleyman Eğitim ve Araştırma Hastanesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cromi A, Ghezzi F, Uccella S, Agosti M, Serati M, Marchitelli G, Bolis P. A randomized trial of preinduction cervical ripening: dinoprostone vaginal insert versus double-balloon catheter. Am J Obstet Gynecol. 2012 Aug;207(2):125.e1-7. doi: 10.1016/j.ajog.2012.05.020. Epub 2012 Jun 1. PMID 22704766
- [Background] Connolly KA, Kohari KS, Rekawek P, Smilen BS, Miller MR, Moshier E, Factor SH, Stone JL, Bianco AT. A randomized trial of Foley balloon induction of labor trial in nulliparas (FIAT-N). Am J Obstet Gynecol. 2016 Sep;215(3):392.e1-6. doi: 10.1016/j.ajog.2016.03.034. Epub 2016 Mar 24. PMID 27018464
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/22704766